CLINICAL TRIAL: NCT00003179
Title: A Two-Part Study of the Treatment of Atypical Endometrial Hyperplasia: Part A: A Prospective Study of Immediate Hysterectomy; Part B: A Randomized Phase II Study of Medroxyprogesterone Acetate Versus Depoprovera
Brief Title: Surgery Plus Medroxyprogesterone in Preventing Endometrial Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: GOG Foundation (Network)
Allocation: Randomized | Purpose: Prevention
Other Study IDs: CDR0000065999; GOG-0167
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-06-10 (Estimated); Status verified 2006-07

CONDITIONS: Endometrial Cancer
Keywords: endometrial cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Medroxyprogesterone

INTERVENTIONS:
Drug: medroxyprogesterone

SUMMARY:
RATIONALE: Chemoprevention therapy is the use of certain drugs to try to prevent the development or recurrence of cancer. The use of surgery with or without medroxyprogesterone may be an effective way to prevent the development of endometrial cancer in patients who have endometrial hyperplasia.

PURPOSE: Phase II trial to compare the effectiveness of surgery alone with that of medroxyprogesterone followed by surgery in preventing endometrial cancer in patients who have endometrial hyperplasia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the joint occurrence of atypical hyperplasia and adenocarcinoma in patients diagnosed at initial biopsy to have complex atypical hyperplasia.
* Compare the histologic response rates in patients with atypical endometrial hyperplasia treated with oral medroxyprogesterone acetate (Provera) vs intramuscular medroxyprogesterone acetate suspension (Depo-Provera) .

OUTLINE: This is a randomized, two-part study.

* Part A: Patients undergo immediate hysterectomy.
* Part B: Patients are randomized to 1 of 2 arms.

  * Arm I: Patients receive oral medroxyprogesterone acetate (Provera) once daily for 3 months.
  * Arm II: Patients receive medroxyprogesterone acetate suspension (Depo- Provera) intramuscularly once monthly for 3 months (days 1, 31, and 62).

Patients undergo hysterectomy at the end of the third month.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A minimum of 360 patients for part A and 140 patients (70 per arm) for part B will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed atypical endometrial hyperplasia with recommended treatment with either:

  * An immediate hysterectomy (Part A) OR
  * A three-month delay prior to hysterectomy and a randomized choice of treatment with oral medroxyprogesterone acetate (Provera) or medroxyprogesterone acetate suspension (Depo-Provera) during the 3 months (Part B with arms I and II)
* Diagnosed by dilation and curettage, Novak curettage, Vabra aspirate or Pipelle endometrial biopsy
* No recognized endometrial carcinoma
* Must not be considered inoperable

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance status:

* GOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 3,000/mm^3
* Platelet count at least 100,000/mm^3
* Granulocyte count at least 1,500/mm^3

Hepatic:

* Bilirubin no greater than 1.5 times normal
* SGOT no greater than 3 times normal
* Alkaline phosphatase no greater than 3 times normal

Renal:

* Creatinine no greater than 2 times normal

Cardiovascular

* No prior thrombophlebitis or thromboembolic phenomena
* No prior cerebrovascular disorders

Other:

* No prior or concurrent malignancy except nonmelanoma skin cancer or carcinoma in situ of the uterine cervix
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* See Disease Characteristics

Radiotherapy:

* Not specified

Surgery:

* See Disease Characteristics

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 1998-11; Primary Completion 2006-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John P. Curtin, MD, Study Chair — Memorial Sloan Kettering Cancer Center; George L. Mutter, MD — Dana-Farber/Brigham and Women's Cancer Center; Francisco A. R. Garcia, MD, MPH — University of Arizona; Richard Zaino, MD — Milton S. Hershey Medical Center
Locations (31):
- United States (30):
  - Arizona Cancer Center, Tucson, Arizona
  - Community Hospital of Los Gatos, Los Gatos, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - Marlene and Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Keesler Medical Center - Keesler AFB, Keesler Air Force Base, Mississippi
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Cooper Hospital/University Medical Center, Camden, New Jersey
  - State University of New York Health Sciences Center - Stony Brook, Stony Brook, New York
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Barrett Cancer Center, Cincinnati, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - University of Oklahoma College of Medicine, Oklahoma City, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Brookview Research, Inc., Nashville, Tennessee
  - University of Texas Medical Branch, Galveston, Texas
  - Fletcher Allen Health Care - Medical Center Campus, Burlington, Vermont
  - Cancer Center at the University of Virginia, Charlottesville, Virginia
- Norwegian Radium Hospital, Oslo, Norway

REFERENCES:
- [Result] Bartels PH, Garcia FA, Trimble CL, Kauderer J, Curtin J, Lim PC, Hess LM, Silverberg S, Zaino RJ, Yozwiak M, Bartels HG, Alberts DS. Karyometry in atypical endometrial hyperplasia: a Gynecologic Oncology Group study. Gynecol Oncol. 2012 Apr;125(1):129-35. doi: 10.1016/j.ygyno.2011.12.422. Epub 2011 Dec 9. PMID 22155796
- [Result] Trimble CL, Kauderer J, Zaino R, Silverberg S, Lim PC, Burke JJ 2nd, Alberts D, Curtin J. Concurrent endometrial carcinoma in women with a biopsy diagnosis of atypical endometrial hyperplasia: a Gynecologic Oncology Group study. Cancer. 2006 Feb 15;106(4):812-9. doi: 10.1002/cncr.21650. PMID 16400639